CLINICAL TRIAL: NCT01495221
Title: To Evaluate The Role of Intravitreal Aflibercept Injection (2.0 mg) in the Management of Previously Treated Patients With Exudative AMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOLD STUDY
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: AMD (With Persistent or Recurrent Fluid Despite Monthly Intravitreal Anti-VEGF Therapy)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal aflibercept (Other): All eligible patients will receive intravitreal aflibercept injection (2.0mg) every 4 weeks (monthly) for the first 12 weeks (3 months), followed by 2 mg once every 8 weeks (2 months) through Week 24. Patients can be dosed as frequently as 2 mg every 4 weeks (monthly) upon investigator discretion.
  Interventions: Drug: Alfilbercept

INTERVENTIONS:
Drug: Alfilbercept — All patients will receive 2.0 mg intravitreal aflibercept injection.

SUMMARY:
This is an open label study to evaluate intravitreally administered 2.0 mg intravitreal aflibercept injection in patients who have been previously treated for AMD and have persistent or recurrent fluid despite monthly intravitreal anti-VEGF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Choroidal neovascularization secondary to AMD
* Best corrected visual acuity in the study eye between 20/25 to 20/400 using an ETDRS chart
* Documentation of presence of subretinal fluid and/or cystoid macular edema on SD-OCT following at least four anti-VEGF treatments within six months before enrollment and a maximum of 5 years of years of treatment for neovascular AMD
* Documentation of presence of subretinal fluid and/or cystoid macular edema less than 30 days since last treatment

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Participation in another simultaneous medical investigation or trial
* Prior treatment with anti-VEGF therapy in the study eye within 30 days of BSL
* Prior treatment with PDT within the past 3 months or more than 4 prior PDT treatments.
* Presence of significant subfoveal fibrosis or atrophy.
* Prior treatment with intravitreal aflibercept injection
* Prior treatment with triamcinolone in the study eye within 6 months of BSL.
* Prior treatment with dexamethasone in the study eye within 30 days prior to BSL
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding BSL
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Ocular or periocular infection
* Active severe intraocular inflammation
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* History of allergy to fluorescein, ICG or iodine, not amenable to treatment
* Known hypersensitivity to aflibercept or to any of the excipients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravitreal Aflibercept
Started | 9 (First Patient enrolled December 2011.)
Completed | 9 (Last patient enrolled May 2012.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 74 [60 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
First Prescription for Choroidial NeoVascularization [Mean (Full Range); unit: Months] | 18.5 [4 to 40]
EDTRS Visual Acuity Score [Mean (Full Range); unit: Letters] | 63 [35 to 79]
Lesion Type: ( Fluroscien Angiogram and [Count of Participants; unit: Participants]
  Occult CNV with PCV features | 3
  Occult CNV with CSC features | 2
  Occult CNV only | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With no Fluid on OCT at Week 24
Description: No primary outcome data can be found or provided.
Time Frame: 24 week
Population: Patients analyzed is zero due to no outcome data was collected at week 24 due to early termination of the clinical study.
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 0

2. Primary Outcome: Mean Change in Visual Acuity From Baseline to Week 16
Description: Visual acuity was documented via BCVA at every study visit.
Time Frame: Baseline to Week 16
Population: The average age of enrollment is 74 years old with first treatment for CNV at 18.5 months.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 9
letters | 4.2 (6.3)

3. Secondary Outcome: Mean Change in OCT Central Retinal Lesion Thickness From Baseline to Week 16
Description: OCT is performed on the Spectralis spectral domain OCT machine (Heidelberg Engineering, Germany). The OCT is centered on the fovea. The OCT examination will use the 19 scan mode on the Spectralis averaging at least 25 images per scan. Follow-up visits will use the follow-up protocol on the Spectralis , automatically placing follow-up scans in precisely the same location as the baseline scan.
Time Frame: Baseline and week 16
Population: The average age of enrollment is 74 years old with first treatment for CNV at 18.5 months.
Measure: Mean (Full Range); unit: Microns
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 9
Microns | -45 [-237 to 237]

4. Secondary Outcome: Mean Change in OCT Greatest Height of Pigment Epithelial Detachment From Baseline to Week 16
Description: as for outcome 3
Time Frame: Baseline and 16 weeks
Population: The average age of enrollment is 74 years old with first treatment for CNV at 18.5 months.
Measure: Mean (Full Range); unit: microns
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 9
microns | -90 [-331 to 331]

ADVERSE EVENTS:
Arm/Group | Intravitreal Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept (N=9)
Left thigh muscle tear and hematoma (Musculoskeletal and connective tissue disorders) | 1 — Not related to treatment
Dog bite to lower left leg (Musculoskeletal and connective tissue disorders) | 1 — Not related to treatment
Unknown Event (General disorders) | 1 — Specific event not documented on patient sheet. Not related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes